CLINICAL TRIAL: NCT02477020
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled, Parallel-group, 6-Week Study to Evaluate the Efficacy and Safety of TAK-063 in Subjects With an Acute Exacerbation of Schizophrenia
Brief Title: A Phase 2 Efficacy and Safety Study of TAK-063 in Participants With an Acute Exacerbation of Schizophrenia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TAK-063-2002; U1111-1169-6472 (Registry Identifier: WHO)
Record Dates: First submitted 2015-06-17; First posted 2015-06-22 (Estimated); Results first posted 2017-09-29 (Actual); Last update posted 2017-09-29 (Actual); Status verified 2017-09

CONDITIONS: Schizophrenia
Keywords: Drug Therapy
MeSH Terms: conditions — Schizophrenia | interventions — 1-(2-fluoro-4-(1H-pyrazol-1-yl)phenyl)-5-methoxy-3-(1-phenyl-1H-pyrazol-5-yl)pyridazin-4(1H)-one

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- TAK-063 20 mg (Experimental): TAK-063 20 mg, tablets, orally, once daily for up to 6 weeks. Dose may be titrated down to 10 mg/day, if intolerable.
  Interventions: Drug: TAK-063 20 mg
- Placebo (Placebo Comparator): TAK-063 matching-placebo tablets, orally, once daily for up to 6 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TAK-063 20 mg — TAK-063 tablet.
  Arms: TAK-063 20 mg
Drug: Placebo — TAK-063 matching-placebo tablet.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy, safety and tolerability of TAK-063 compared with placebo in treatment of acutely exacerbated schizophrenia.

DETAILED DESCRIPTION:
The drug being tested in this study is called TAK-063. TAK-063 is being tested to treat people who have schizophrenia. This study will look at the different symptoms associated with schizophrenia including cognitive symptoms, personal and social functioning and functional capacity (ability to perform tasks associated with real, everyday life such as household chores, communication, finance, transportation, and planning recreational activities) in people who take TAK-063.

The study enrolled 164 patients. Participants were randomly assigned (by chance, like flipping a coin) to one of the two treatment groups-which will remain undisclosed to the patient and study doctor during the study (unless there is an urgent medical need):

* TAK-063 20 mg
* Placebo (dummy inactive pill) - this is a tablet that looks like the study drug but has no active ingredient.

All participants will be asked to take the tablets once daily at nighttime. All participants will initially receive TAK-063, 20 mg/day. The dose may be titrated down to 10 mg/day, if intolerable.

The multi-center trial will be conducted in the United States. The overall time to participate in this study is 6 weeks. Participants will be hospitalized until the Week 3 visit. Participants will make 11 visits to the clinic during the treatment and 1 visit during the follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Is capable of understanding and complying with protocol requirements.
2. The participants or, when applicable, the participant's legally acceptable representative signs and dates a written, informed consent form and any required privacy authorization prior to the initiation of any study procedures.
3. Has a primary diagnosis of schizophrenia (Diagnostic and Statistical Manual of Mental Disorders, 5th Edition [DSM-5], 295.90) confirmed by clinical interview (Structured Clinical Interview for DSM-5 Clinical Trial Version [SCID-5-CT]). The participant's initial diagnosis must be greater than or equal to (>=) 1 year from screening.
4. Is a man or woman age 18 to 65, inclusive, at Screening.
5. Male participant who is nonsterilized and sexually active with a female partner of child bearing potential agrees to use adequate contraception from signing of informed consent throughout the duration of the study and for 12 weeks after last dose.
6. Female participant of childbearing potential who is sexually active with a nonsterilized male partner agrees to use adequate contraception from signing of informed consent throughout the duration of the study and for 12 weeks after last dose.
7. The participant's psychotic symptoms were exacerbated within 2 months (60 days) prior to Screening (example, aggravated delusion).
8. Has a score of 5 (moderate severe) or higher in 3 or more items of the following Positive and Negative Symptom Scale (PANSS) items at Screening and Day 1: delusions (P1), conceptual disorganization (P2), hallucinations (P3), suspiciousness (P6), and unusual thought content (G9).
9. Has a PANSS total score of 80 or higher at Screening and Day 1.
10. Has a Clinical Global Impression Scale- Severity of Illness Scale (CGI-S) of 4 or greater at Screening and Day 1.
11. Is able and agrees to remain off prior antipsychotic medication and all excluded medications as outlined in the protocol for the duration of the study.
12. Has an identified, reliable caregiver. A caregiver is defined as a family member, informant or friend who is able and willing to assist and support the administration of study drug, adherence to protocol requirements and to the study schedule.
13. Has a body mass index (BMI) score between 18.0 and 35.0 kilogram per square meter (kg/m^2), inclusive, at Screening.

Exclusion Criteria:

1. Has received any investigational compound within 30 days prior to Screening, or within 5 half-lives prior to screening, whichever is longer.
2. Has received TAK-063 in a previous clinical study or as a therapeutic agent or has previously or is currently participating in this study or have participated in 2 or more clinical studies within 12 months prior to Screening.
3. Has a decrease in the PANSS Total Score by 20 percent (%) or more at Baseline (Day 1) compared with that at Screening [(PANSS Total Score at Screening- PANSS total score at Baseline)/(PANSS Total Score at Screening- 30)]*100 >=20%].
4. Is an immediate family member, study site employee, or in a dependent relationship with a study site employee who is involved in the conduct of this study (example, spouse, parent, child, and sibling) or may consent under duress.
5. Has uncontrolled, clinically significant neurologic, cardiovascular, pulmonary, hepatic, renal, metabolic, gastrointestinal, or endocrine disease or other abnormality (other than the disease being studied), which may impact the ability of the participant to participate or potentially confound the study results.
6. Has a history of severe head injury/traumatic brain injury, myocardial infarction or stroke.
7. Has a known hypersensitivity to any component of the formulation of TAK-063 or the practice pills (i.e., small colored candies) during the AiCure device training.
8. Has a positive urine drug result (illicit, illegal or without valid prescription or medical need) at Screening.
9. Has a moderate or severe substance use disorder (meeting more than 5 diagnostic criteria of DSM-5 either currently or within the last 6 months) for alcohol or other substances of abuse except nicotine or caffeine.
10. Has taken any excluded medication, supplements, or food products or has had insufficient washout of medications, supplements, or food products as listed in the Excluded /Allowed Medications, Procedures, and Treatments table or is unable or unwilling to discontinue medications as required by the protocol.
11. If female, the participant is pregnant or lactating or intending to become pregnant (a positive pregnancy test at Screening or Day 1), or intending to donate ova, before or during the course of the study or within 12 weeks after last dose.
12. If male, the participant intends to donate sperm during the course of this study or for 12 weeks after last dose.
13. Has a psychiatric disorder other than schizophrenia as their primary diagnosis.
14. Has a history of or known personality disorder or other psychiatric disorder that, in the opinion of the investigator, would interfere with participation in the study.
15. Has a history of neuroleptic malignant syndrome, water intoxication, or paralytic ileus or other conditions that may interfere with absorption of study medication.
16. Is considered by the investigator to be at imminent risk of suicide or injury to self, others, or property or participants who within the past year prior to Screening have attempted suicide or have positive answers on item 4 or 5 on the Columbia Suicide Severity Rating Scale (C-SSRS) at Screening or Day 1.
17. Has Parkinson disease, tardive dyskinesia, or other chronic movement disorder that may interfere with the interpretation of study results.
18. Has any existing or previous history of cancer that has been in remission for less than 5 years prior to Screening. (This criterion does not include those participants with basal cell, stage I squamous cell skin cancer or in situ cervical cancer).
19. Has newly diagnosed diabetes or requiring insulin for their treatment; diabetic participants that have had changes to their diabetic treatment regimen within 30 days prior to screening or diabetic participants that have had hospitalizations for their diabetes and/or diabetes related conditions in the past year prior to screening.
20. Has long QT syndrome or under the treatment with Class 1A (example, quinidine, procainamide) or Class 3 (example, amiodarone, sotalol) anti-arrhythmic drugs.
21. Is known to be currently infected or have been infected with human immunodeficiency virus (HIV), hepatitis B virus (HBV), or hepatitis C virus (HCV).
22. Has received any depot preparation (sustained-release formulation) of antipsychotic drugs within 1 month (30 days) of Screening.
23. Has received clozapine for the treatment of schizophrenia (lifetime) before screening (this does not include the use of low-dose clozapine for sleep).
24. Has received monoamine oxidase (MAO) inhibitors or fluoxetine within 1 month (30 days) before Screening.
25. Is considered to be treatment resistant. Treatment resistance is defined as prior nonresponse to 2 courses of treatment with antipsychotics of different chemical classes for at least 4 weeks each at doses considered to be effective.
26. Has received electroconvulsive therapy within 6 months (180 days) before Screening.
27. Has a history of hypersensitivity to more than one distinct chemical class of drug (including anaphylaxis, rash, or urticaria caused by drugs).
28. Is considered otherwise inappropriate for the study by the investigator or Sponsor's medical monitor and/or designee.
29. Has 1 or more laboratory values outside the normal range that are considered by the investigator to be clinically significant at the Screening Visit; or has any of the following at the Screening Visit: a serum creatinine value >1.5 times the upper limit of normal (ULN). A total serum total bilirubin value >1.5*ULN. A serum alanine aminotransferase (ALT) or aspartate aminotransferase (AST) value >2*ULN, or prolactin >= 100 nanogram/milliliter (ng/mL).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 2015-07-01 (Actual); Primary Completion 2016-07-13 (Actual); Study Completion 2016-07-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda
Locations (15):
- United States (15):
  - Springdale, Alaska
  - Culver City, California
  - Lemon Grove, California
  - Long Beach, California
  - Pico Rivera, California
  - Lauderhill, Florida
  - Orlando, Florida
  - Atlanta, Georgia
  - Lake Charles, Louisiana
  - St Louis, Missouri
  - Las Vegas, Nevada
  - Oklahoma City, Oklahoma
  - Austin, Texas
  - Dallas, Texas
  - Houston, Texas

REFERENCES:
- [Derived] Macek TA, McCue M, Dong X, Hanson E, Goldsmith P, Affinito J, Mahableshwarkar AR. A phase 2, randomized, placebo-controlled study of the efficacy and safety of TAK-063 in subjects with an acute exacerbation of schizophrenia. Schizophr Res. 2019 Feb;204:289-294. doi: 10.1016/j.schres.2018.08.028. Epub 2018 Sep 3. PMID 30190165
- [Derived] Tohyama K, Sudo M, Morohashi A, Kato S, Takahashi J, Tagawa Y. Pre-clinical Characterization of Absorption, Distribution, Metabolism and Excretion Properties of TAK-063. Basic Clin Pharmacol Toxicol. 2018 Jun;122(6):577-587. doi: 10.1111/bcpt.12964. Epub 2018 Feb 26. PMID 29345044

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 13 investigative sites in United States from 01 July 2015 to 27 July 2016.
Pre-assignment Details: Participants with a diagnosis of acute exacerbation of schizophrenia were enrolled in two treatment groups TAK-063 or placebo.
Groups:
- TAK-063: TAK-063 20 mg, tablets, orally, once daily for up to 6 weeks.
Period: Overall Study
Arm/Group | Placebo | TAK-063
Started | 81 | 83
Completed | 51 (Completed = participants who completed study treatment.) | 55 (Completed = participants who completed study treatment.)
Not Completed | 30 | 28
Not completed — Pretreatment Event/Adverse Event | 6 | 6
Not completed — Voluntary Withdrawal | 7 | 16
Not completed — Reason not Specified | 3 | 1
Not completed — Lack of Efficacy | 14 | 5

BASELINE CHARACTERISTICS:
Population: All randomized participants who received at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | TAK-063 | Total
Number analyzed (Participants) | 81 | 83 | 164
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.2 (10.44) | 42.3 (10.36) | 41.8 (10.38)
Age, Customized [Number; unit: participants]
  18 - 50 years | 62 | 57 | 119
  51 - 65 years | 19 | 26 | 45
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 18 | 32
  Male | 67 | 65 | 132
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 14 | 6 | 20
  Non-Hispanic and Latino | 67 | 77 | 144
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Black or African American | 43 | 65 | 108
  White | 33 | 16 | 49
  Multiracial | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 81 | 83 | 164
Height [Mean (Standard Deviation); unit: cm] | 176.1 (9.02) | 174.3 (9.41) | 175.2 (9.23)
Weight [Mean (Standard Deviation); unit: kg] | 86.64 (16.490) | 82.46 (15.480) | 84.52 (16.075)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — BMI = Weight (kg)/height (m^2)
  kg/m^2 | 27.84 (4.427) | 27.17 (4.231) | 27.50 (4.329)
Smoking Classification [Number; unit: participants]
  Has never smoked | 7 | 7 | 14
  Is a current smoker | 67 | 73 | 140
  Is an ex-smoker | 7 | 3 | 10
Alcohol Classification [Number; unit: participants]
  Has never drunk | 27 | 21 | 48
  Is a current drinker | 21 | 31 | 52
  Is an ex-drinker | 33 | 31 | 64
Consume Caffeine [Number; unit: participants]
  Yes | 73 | 74 | 147
  No | 8 | 9 | 17
Female Reproductive Status [Number; unit: participants]
  Postmenopausal | 7 | 4 | 11
  Surgically Sterile | 1 | 6 | 7
  Female of Childbearing Potential | 6 | 8 | 14
  Not applicable (Male participant) | 67 | 65 | 132

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Positive and Negative Symptom Scale (PANSS) Total Score at Week 6
Description: PANSS assesses the positive symptoms, negative symptoms, and general psychopathology specifically associated with schizophrenia. The scale consists of 30 items. Each item is rated on a scale from 1 (symptom not present) to 7 (symptoms extremely severe). The sum of the 30 items is defined as the PANSS total score and ranges from 30 to 210; higher score indicates greater severity. Least square mean and standard error values were determined using a mixed model for repeated measures (MMRM). A negative change from Baseline indicates improvement.
Time Frame: Baseline and Week 6
Population: The full analysis set included all participants who were randomized, received at least one dose of study drug and have a baseline value and at least one valid postbaseline value for assessment of primary efficacy. Here number of participants analyzed are participants evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | TAK-063
Number analyzed (Participants) | 51 | 55
score on a scale | -14.08 (2.474) | -19.54 (2.412)
Statistical Analysis 1: Comparison: Placebo vs TAK-063; Test type: Superiority or Other; p = 0.115, MMRM — No adjustment for multiple comparisons. Least square means, differences and p-values were obtained using MMRM; Least square mean difference = -5.46, 95% CI 2-sided [-12.26 to 1.35], Standard Error of Mean 3.442 — TAK-063 - Placebo. Baseline Positive and Negative Symptom Scale (PANSS) total score was used as covariate, pooled center, week and treatment as fixed factors, treatment-by-week interaction and Baseline PANSS total score-by-week interaction

2. Secondary Outcome: Change From Baseline in PANSS Total Score at Weeks 1, 2, 3, 4 and 5
Description: PANSS assesses the positive symptoms, negative symptoms, and general psychopathology specifically associated with schizophrenia. The scale consists of 30 items. Each item is rated on a scale from 1 (symptom not present) to 7 (symptoms extremely severe). The sum of the 30 items is defined as the PANSS total score and ranges from 30 to 210; higher score indicates greater severity. Least square mean and standard error values were determined using a MMRM. A negative change from Baseline indicates improvement.
Time Frame: Baseline and Weeks 1, 2, 3, 4 and 5
Population: The full analysis set included all participants who were randomized, received at least one dose of study drug and have a baseline value and at least one valid postbaseline value for assessment of primary efficacy. Here 'n' refers to number of participants analyzed at each time point.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | TAK-063
Number analyzed (Participants) | 76 | 80
score on a scale
  Change at Week 1 (n = 76, 80) | -8.30 (1.106) | -9.09 (1.075)
  Change at Week 2 (n = 72, 72) | -9.73 (1.604) | -11.95 (1.580)
  Change at Week 3 (n = 67, 68) | -10.91 (2.017) | -14.37 (1.985)
  Change at Week 4 (n = 57, 60) | -12.80 (2.256) | -14.91 (2.212)
  Change at Week 5 (n = 53, 58) | -13.03 (2.321) | -16.94 (2.268)
Statistical Analysis 1: Comparison: Placebo vs TAK-063; Change at Week 1; Test type: Superiority or Other; p = 0.602, MMRM — No adjustment for multiple comparisons. Least square means, differences and p-values were obtained using MMRM; Least square mean difference = -0.79, 95% CI 2-sided [-3.77 to 2.19], Standard Error of Mean 1.508 — TAK-063 - Placebo. Baseline PANSS total score was used as covariate, pooled center, week and treatment as fixed factors, treatment-by-week interaction and Baseline PANSS total score-by-week interaction
Statistical Analysis 2: Comparison: Placebo vs TAK-063; Change at Week 2; Test type: Superiority or Other; p = 0.322, MMRM — No adjustment for multiple comparisons. Least square means, differences and p-values were obtained using a MMRM; Least square mean difference = -2.22, 95% CI 2-sided [-6.62 to 2.19], Standard Error of Mean 2.229 — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs TAK-063; Change at Week 3; Test type: Superiority or Other; p = 0.221, MMRM — No adjustment for multiple comparisons. Least square means, differences and p-values were obtained using a MMRM; Least square mean difference = -3.46, 95% CI 2-sided [-9.02 to 2.10], Standard Error of Mean 2.813 — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 4: Comparison: Placebo vs TAK-063; Change at Week 4; Test type: Superiority or Other; p = 0.504, MMRM — No adjustment for multiple comparisons. Least square means, differences and p-values were obtained using a MMRM; Least square mean difference = -2.11, 95% CI 2-sided [-8.33 to 4.11], Standard Error of Mean 3.147 — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 5: Comparison: Placebo vs TAK-063; Change at Week 5; Test type: Superiority or Other; p = 0.229, MMRM — No adjustment for multiple comparisons. Least square means, differences and p-values were obtained using a MMRM; Least square mean difference = -3.91, 95% CI 2-sided [-10.30 to 2.48], Standard Error of Mean 3.231 — [estimate comment as in outcome 2, analysis 1]

3. Secondary Outcome: Change From Baseline in PANSS Subscales Using the Marder 5-factor Model at Weeks 1, 2, 3, 4, 5, and 6
Description: PANSS subscales using the Marder 5-factor model include positive symptoms (8-items, total score = total score = 8 to 56, with a higher score indicating greater severity of symptoms), negative symptoms (7-items, total score = 7 to 49, with a higher score indicating greater severity of symptoms), disorganized thoughts (7-items, total score = 7 to 49, with a higher score indicating greater severity of symptoms), impulsivity/hostility (4-items, total score = 4 to 28, with a higher score indicating greater severity of symptoms), anxiety/depression (4-items, total score = 4 to 28, with a higher score indicating greater severity of symptoms). Responses to each item range from 1 = absence of symptom, to 7 = most extreme symptoms. An improvement in symptoms is represented by change from baseline values that are negative.
Time Frame: Baseline and Weeks 1, 2, 3, 4, 5 and 6
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | TAK-063
Number analyzed (Participants) | 76 | 80
score on a scale
  Positive symptoms, Change at Week 1 (n=76,80) | -2.64 (0.410) | -3.37 (0.397)
  Positive symptoms, Change at Week 2 (n=72,72) | -3.20 (0.561) | -4.39 (0.554)
  Positive symptoms, Change at Week 3 (n=67,68) | -3.67 (0.683) | -5.61 (0.674)
  Positive symptoms, Change at Week 4 (n=57,60) | -4.49 (0.731) | -6.03 (0.717)
  Positive symptoms, Change at Week 5 (n=53,58) | -4.65 (0.779) | -6.67 (0.760)
  Positive symptoms, Change at Week 6 (n=51,55) | -5.33 (0.800) | -7.23 (0.778)
  Negative symptoms, Change at Week 1 (n=76,80) | -1.67 (0.415) | -1.33 (0.405)
  Negative symptoms, Change at Week 2 (n=72,72) | -1.88 (0.545) | -2.49 (0.538)
  Negative symptoms, Change at Week 3 (n=67,68) | -2.87 (0.589) | -2.72 (0.580)
  Negative symptoms, Change at Week 4 (n=57,60) | -2.64 (0.673) | -3.23 (0.661)
  Negative symptoms, Change at Week 5 (n=53,58) | -3.01 (0.679) | -3.15 (0.662)
  Negative symptoms, Change at Week 6 (n=51,55) | -3.38 (0.681) | -4.11 (0.662)
  Disorganized thoughts, Change at Week 1 (n=76,80) | -1.04 (0.298) | -1.41 (0.290)
  Disorganized thoughts, Change at Week 2 (n=72,72) | -1.55 (0.382) | -1.77 (0.377)
  Disorganized thoughts, Change at Week 3 (n=67,68) | -1.60 (0.444) | -2.06 (0.439)
  Disorganized thoughts, Change at Week 4 (n=57,60) | -1.92 (0.505) | -1.92 (0.497)
  Disorganized thoughts, Change at Week 5 (n=53,58) | -1.37 (0.562) | -2.10 (0.550)
  Disorganized thoughts, Change at Week 6 (n=51,55) | -1.90 (0.579) | -3.16 (0.565)
  Hostility, Change at Week 1 (n=76,80) | -1.32 (0.342) | -1.64 (0.334)
  Hostility, Change at Week 2 (n=72,72) | -1.40 (0.364) | -1.36 (0.360)
  Hostility, Change at Week 3 (n=67,68) | -0.83 (0.434) | -1.70 (0.430)
  Hostility, Change at Week 4 (n=57,60) | -1.21 (0.492) | -1.21 (0.482)
  Hostility, Change at Week 5 (n=53,58) | -1.43 (0.494) | -2.04 (0.478)
  Hostility, Change at Week 6 (n=51,55) | -1.16 (0.476) | -2.28 (0.462)
  Anxiety, Change at Week 1 (n=76,80) | -2.11 (0.290) | -1.86 (0.284)
  Anxiety, Change at Week 2 (n=72,72) | -2.29 (0.361) | -2.70 (0.359)
  Anxiety, Change at Week 3 (n=67,68) | -2.70 (0.376) | -3.19 (0.373)
  Anxiety, Change at Week 4 (n=57,60) | -3.42 (0.427) | -3.74 (0.419)
  Anxiety, Change at Week 5 (n=53,58) | -3.80 (0.414) | -4.32 (0.402)
  Anxiety, Change at Week 6 (n=51,55) | -3.66 (0.460) | -4.34 (0.447)
Statistical Analysis 1: Comparison: Placebo vs TAK-063; Positive symptoms, Change at Week 1; Test type: Superiority or Other; p = 0.195, MMRM — No adjustment for multiple comparisons. Least square means, differences and p-values were obtained using a MMRM; Least square mean difference = -0.73, 95% CI 2-sided [-1.84 to 0.38], Standard Error of Mean 0.562 — TAK-063 - Placebo. PANSS Marder five-factor score was used as a covariate, pooled center, week and treatment as fixed factors, the treatment-by-week interaction, and Baseline PANSS Marder five-factor score-by-week interaction
Statistical Analysis 2: Comparison: Placebo vs TAK-063; Positive symptoms, Change at Week 2; Test type: Superiority or Other; p = 0.132, MMRM — No adjustment for multiple comparisons. Least square means, differences and p-values were obtained using a MMRM; Least square mean difference = -1.19, 95% CI 2-sided [-2.74 to 0.36], Standard Error of Mean 0.786 — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs TAK-063; Positive symptoms, Change at Week 3; Test type: Superiority or Other; p = 0.045, MMRM — No adjustment for multiple comparisons. Least square means, differences and p-values were obtained using a MMRM; Least square mean difference = -1.94, 95% CI 2-sided [-3.84 to -0.05], Standard Error of Mean 0.959 — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 4: Comparison: Placebo vs TAK-063; Positive symptoms, Change at Week 4; Test type: Superiority or Other; p = 0.135, MMRM — No adjustment for multiple comparisons. Least square means, differences and p-values were obtained using a MMRM; Least square mean difference = -1.54, 95% CI 2-sided [-3.56 to 0.49], Standard Error of Mean 1.025 — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 5: Comparison: Placebo vs TAK-063; Positive symptoms, Change at Week 5; Test type: Superiority or Other; p = 0.067, MMRM — No adjustment for multiple comparisons. Least square means, differences and p-values were obtained using a MMRM; Least square mean difference = -2.01, 95% CI 2-sided [-4.17 to 0.14], Standard Error of Mean 1.090 — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 6: Comparison: Placebo vs TAK-063; Positive symptoms, Change at Week 6; Test type: Superiority or Other; p = 0.092, MMRM — No adjustment for multiple comparisons. Least square means, differences and p-values were obtained using a MMRM; Least square mean difference = -1.90, 95% CI 2-sided [-4.11 to 0.31], Standard Error of Mean 1.119 — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 7: Comparison: Placebo vs TAK-063; Negative symptoms, Change at Week 1; Test type: Superiority or Other; p = 0.548, MMRM — No adjustment for multiple comparisons. Least square means, differences and p-values were obtained using a MMRM; Least square mean difference = 0.34, 95% CI 2-sided [-0.78 to 1.46], Standard Error of Mean 0.566 — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 8: Comparison: Placebo vs TAK-063; Negative symptoms, Change at Week 2; Test type: Superiority or Other; p = 0.420, MMRM — No adjustment for multiple comparisons. Least square means, differences and p-values were obtained using a MMRM; Least square mean difference = -0.61, 95% CI 2-sided [-2.11 to 0.88], Standard Error of Mean 0.756 — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 9: Comparison: Placebo vs TAK-063; Negative symptoms, Change at Week 3; Test type: Superiority or Other; p = 0.857, MMRM — No adjustment for multiple comparisons. Least square means, differences and p-values were obtained using a MMRM; Least square mean difference = 0.15, 95% CI 2-sided [-1.47 to 1.76], Standard Error of Mean 0.818 — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 10: Comparison: Placebo vs TAK-063; Negative symptoms, Change at Week 4; Test type: Superiority or Other; p = 0.527, MMRM — No adjustment for multiple comparisons. Least square means, differences and p-values were obtained using a MMRM; Least square mean difference = -0.59, 95% CI 2-sided [-2.44 to 1.26], Standard Error of Mean 0.936 — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 11: Comparison: Placebo vs TAK-063; Negative symptoms, Change at Week 5; Test type: Superiority or Other; p = 0.875, MMRM — No adjustment for multiple comparisons. Least square means, differences and p-values were obtained using a MMRM; Least square mean difference = -0.15, 95% CI 2-sided [-2.01 to 1.71], Standard Error of Mean 0.940 — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 12: Comparison: Placebo vs TAK-063; Negative symptoms, Change at Week 6; Test type: Superiority or Other; p = 0.441, MMRM — No adjustment for multiple comparisons. Least square means, differences and p-values were obtained using a MMRM; Least square mean difference = -0.73, 95% CI 2-sided [-2.58 to 1.13], Standard Error of Mean 0.940 — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 13: Comparison: Placebo vs TAK-063; Disorganized thoughts, Change at Week 1; Test type: Superiority or Other; p = 0.362, MMRM — No adjustment for multiple comparisons. Least square means, differences and p-values were obtained using a MMRM; Least square mean difference = -0.37, 95% CI 2-sided [-1.17 to 0.43], Standard Error of Mean 0.406 — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 14: Comparison: Placebo vs TAK-063; Disorganized thoughts, Change at Week 2; Test type: Superiority or Other; p = 0.687, MMRM — No adjustment for multiple comparisons. Least square means, differences and p-values were obtained using a MMRM; Least square mean difference = -0.21, 95% CI 2-sided [-1.26 to 0.83], Standard Error of Mean 0.530 — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 15: Comparison: Placebo vs TAK-063; Disorganized thoughts, Change at Week 3; Test type: Superiority or Other; p = 0.458, MMRM — No adjustment for multiple comparisons. Least square means, differences and p-values were obtained using a MMRM; Least square mean difference = -0.46, 95% CI 2-sided [-1.68 to 0.76], Standard Error of Mean 0.618 — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 16: Comparison: Placebo vs TAK-063; Disorganized thoughts, Change at Week 4; Test type: Superiority or Other; p = 0.991, MMRM — No adjustment for multiple comparisons. Least square means, differences and p-values were obtained using a MMRM; Least square mean difference = 0.01, 95% CI 2-sided [-1.38 to 1.40], Standard Error of Mean 0.704 — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 17: Comparison: Placebo vs TAK-063; Disorganized thoughts, Change at Week 5; Test type: Superiority or Other; p = 0.354, MMRM — No adjustment for multiple comparisons. Least square means, differences and p-values were obtained using a MMRM; Least square mean difference = -0.73, 95% CI 2-sided [-2.27 to 0.82], Standard Error of Mean 0.782 — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 18: Comparison: Placebo vs TAK-063; Disorganized thoughts, Change at Week 6; Test type: Superiority or Other; p = 0.119, MMRM — No adjustment for multiple comparisons. Least square means, differences and p-values were obtained using a MMRM; Least square mean difference = -1.26, 95% CI 2-sided [-2.85 to 0.33], Standard Error of Mean 0.804 — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 19: Comparison: Placebo vs TAK-063; Hostility, Change at Week 1; Test type: Superiority or Other; p = 0.493, MMRM — No adjustment for multiple comparisons. Least square means, differences and p-values were obtained using a MMRM; Least square mean difference = -0.32, 95% CI 2-sided [-1.25 to 0.60], Standard Error of Mean 0.469 — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 20: Comparison: Placebo vs TAK-063; Hostility, Change at Week 2; Test type: Superiority or Other; p = 0.949, MMRM — No adjustment for multiple comparisons. Least square means, differences and p-values were obtained using a MMRM; Least square mean difference = 0.03, 95% CI 2-sided [-0.96 to 1.03], Standard Error of Mean 0.504 — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 21: Comparison: Placebo vs TAK-063; Hostility, Change at Week 3; Test type: Superiority or Other; p = 0.153, MMRM — No adjustment for multiple comparisons. Least square means, differences and p-values were obtained using a MMRM; Least square mean difference = -0.87, 95% CI 2-sided [-2.06 to 0.33], Standard Error of Mean 0.604 — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 22: Comparison: Placebo vs TAK-063; Hostility, Change at Week 4; Test type: Superiority or Other; p = 0.994, MMRM — No adjustment for multiple comparisons. Least square means, differences and p-values were obtained using a MMRM; Least square mean difference = 0.00, 95% CI 2-sided [-1.34 to 1.35], Standard Error of Mean 0.681 — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 23: Comparison: Placebo vs TAK-063; Hostility, Change at Week 5; Test type: Superiority or Other; p = 0.365, MMRM — No adjustment for multiple comparisons. Least square means, differences and p-values were obtained using a MMRM; Least square mean difference = -0.62, 95% CI 2-sided [-1.96 to 0.73], Standard Error of Mean 0.679 — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 24: Comparison: Placebo vs TAK-063; Hostility, Change at Week 6; Test type: Superiority or Other; p = 0.088, MMRM — No adjustment for multiple comparisons. Least square means, differences and p-values were obtained using a MMRM; Least square mean difference = -1.12, 95% CI 2-sided [-2.41 to 0.17], Standard Error of Mean 0.653 — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 25: Comparison: Placebo vs TAK-063; Anxiety, Change at Week 1; Test type: Superiority or Other; p = 0.535, MMRM — No adjustment for multiple comparisons. Least square means, differences and p-values were obtained using a MMRM; Least square mean difference = 0.25, 95% CI 2-sided [-0.54 to 1.03], Standard Error of Mean 0.397 — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 26: Comparison: Placebo vs TAK-063; Anxiety, Change at Week 2; Test type: Superiority or Other; p = 0.412, MMRM — No adjustment for multiple comparisons. Least square means, differences and p-values were obtained using a MMRM; Least square mean difference = -0.41, 95% CI 2-sided [-1.40 to 0.58], Standard Error of Mean 0.502 — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 27: Comparison: Placebo vs TAK-063; Anxiety, Change at Week 3; Test type: Superiority or Other; p = 0.354, MMRM — No adjustment for multiple comparisons. Least square means, differences and p-values were obtained using a MMRM; Least square mean difference = -0.49, 95% CI 2-sided [-1.52 to 0.55], Standard Error of Mean 0.522 — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 28: Comparison: Placebo vs TAK-063; Anxiety, Change at Week 4; Test type: Superiority or Other; p = 0.589, MMRM — No adjustment for multiple comparisons. Least square means, differences and p-values were obtained using a MMRM; Least square mean difference = -0.32, 95% CI 2-sided [-1.49 to 0.85], Standard Error of Mean 0.590 — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 29: Comparison: Placebo vs TAK-063; Anxiety, Change at Week 5; Test type: Superiority or Other; p = 0.360, MMRM — No adjustment for multiple comparisons. Least square means, differences and p-values were obtained using a MMRM; Least square mean difference = -0.52, 95% CI 2-sided [-1.65 to 0.60], Standard Error of Mean 0.569 — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 30: Comparison: Placebo vs TAK-063; Anxiety, Change at Week 6; Test type: Superiority or Other; p = 0.288, MMRM — No adjustment for multiple comparisons. Least square means, differences and p-values were obtained using a MMRM; Least square mean difference = -0.68, 95% CI 2-sided [-1.93 to 0.58], Standard Error of Mean 0.635 — [estimate comment as in outcome 3, analysis 1]

4. Secondary Outcome: Change From Baseline in PANSS Subscales at Weeks 1, 2, 3, 4, 5 and 6
Description: PANSS assesses the positive symptoms, negative symptoms, and general psychopathology specifically associated with schizophrenia. The scale consists of 30 items. Each item is rated on a scale from 1 (symptom not present) to 7 (symptoms extremely severe). Positive subscale consists of 7 items which assesses the positive symptoms with subscale score ranging from 7 to 49, where higher score indicates greater severity. Negative subscale consists of 7 items which assesses the negative symptoms with subscale score ranging from 7 to 49, where higher score indicates greater severity. General psychopathology subscale consists of 16 items which assesses the general symptoms of schizophrenia with subscale score ranging from 16 to 96, where higher score indicates greater severity. Least square mean and standard error values were determined using a MMRM. A negative change from Baseline indicates improvement.
Time Frame: Baseline and Weeks 1, 2, 3, 4, 5 and 6
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | TAK-063
Number analyzed (Participants) | 76 | 80
score on a scale
  PANSS Positive Score, Change at Week 1 (n=76,80) | -2.80 (0.434) | -3.49 (0.420)
  PANSS Positive Score, Change at Week 2 (n=72,72) | -3.63 (0.566) | -4.35 (0.556)
  PANSS Positive Score, Change at Week 3 (n=67,68) | -3.87 (0.677) | -5.35 (0.666)
  PANSS Positive Score, Change at Week 4 (n=57,60) | -4.42 (0.729) | -5.62 (0.715)
  PANSS Positive Score, Change at Week 5 (n=53,58) | -4.61 (0.757) | -6.33 (0.738)
  PANSS Positive Score, Change at Week 6 (n=51,55) | -5.35 (0.789) | -6.95 (0.767)
  PANSS Negative Score, Change at Week 1 (n=76,80) | -1.30 (0.369) | -1.24 (0.360)
  PANSS Negative Score, Change at Week 2 (n=72,72) | -1.12 (0.498) | -1.71 (0.493)
  PANSS Negative Score, Change at Week 3 (n=67,68) | -1.77 (0.519) | -2.14 (0.513)
  PANSS Negative Score, Change at Week 4 (n=57,60) | -1.98 (0.615) | -2.35 (0.604)
  PANSS Negative Score, Change at Week 5 (n=53,58) | -2.14 (0.644) | -2.36 (0.627)
  PANSS Negative Score, Change at Week 6 (n=51,55) | -2.29 (0.617) | -3.44 (0.599)
  PANSS General Score, Change at Week 1 (n=76,80) | -4.54 (0.587) | -4.47 (0.573)
  PANSS General Score, Change at Week 2 (n=72,72) | -5.43 (0.828) | -6.05 (0.819)
  PANSS General Score, Change at Week 3 (n=67,68) | -5.85 (1.043) | -7.15 (1.029)
  PANSS General Score, Change at Week 4 (n=57,60) | -6.96 (1.165) | -7.33 (1.146)
  PANSS General Score, Change at Week 5 (n=53,58) | -7.12 (1.166) | -8.73 (1.140)
  PANSS General Score, Change at Week 6 (n=51,55) | -7.35 (1.245) | -9.79 (1.217)
Statistical Analysis 1: Comparison: Placebo vs TAK-063; PANSS Positive Score, Change at Week 1; Test type: Superiority or Other; p = 0.238, MMRM — No adjustment for multiple comparisons. Least square means, differences and p-values were obtained using a MMRM; Least square mean difference = -0.70, 95% CI 2-sided [-1.87 to 0.47], Standard Error of Mean 0.590 — TAK-063 - Placebo. PANSS subscale score was used as a covariate, pooled center, week and treatment as fixed factors, the treatment-by-week interaction and Baseline PANSS subscale score-by-week interaction
Statistical Analysis 2: Comparison: Placebo vs TAK-063; PANSS Positive Score, Change at Week 2; Test type: Superiority or Other; p = 0.359, MMRM — No adjustment for multiple comparisons. Least square means, differences and p-values were obtained using a MMRM; Least square mean difference = -0.72, 95% CI 2-sided [-2.27 to 0.83], Standard Error of Mean 0.784 — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs TAK-063; PANSS Positive Score, Change at Week 3; Test type: Superiority or Other; p = 0.119, MMRM — No adjustment for multiple comparisons. Least square means, differences and p-values were obtained using a MMRM; Least square mean difference = -1.48, 95% CI 2-sided [-3.34 to 0.38], Standard Error of Mean 0.943 — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 4: Comparison: Placebo vs TAK-063; PANSS Positive Score, Change at Week 4; Test type: Superiority or Other; p = 0.238, MMRM — No adjustment for multiple comparisons. Least square means, differences and p-values were obtained using a MMRM; Least square mean difference = -1.20, 95% CI 2-sided [-3.21 to 0.80], Standard Error of Mean 1.014 — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 5: Comparison: Placebo vs TAK-063; PANSS Positive Score, Change at Week 5; Test type: Superiority or Other; p = 0.102, MMRM — No adjustment for multiple comparisons. Least square means, differences and p-values were obtained using a MMRM; Least square mean difference = -1.73, 95% CI 2-sided [-3.81 to 0.35], Standard Error of Mean 1.051 — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 6: Comparison: Placebo vs TAK-063; PANSS Positive Score, Change at Week 6; Test type: Superiority or Other; p = 0.145, MMRM — No adjustment for multiple comparisons. Least square means, differences and p-values were obtained using a MMRM; Least square mean difference = -1.60, 95% CI 2-sided [-3.77 to 0.56], Standard Error of Mean 1.094 — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 7: Comparison: Placebo vs TAK-063; PANSS Negative Score, Change at Week 1; Test type: Superiority or Other; p = 0.902, MMRM — No adjustment for multiple comparisons. Least square means, differences and p-values were obtained using a MMRM; Least square mean difference = 0.06, 95% CI 2-sided [-0.93 to 1.06], Standard Error of Mean 0.504 — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 8: Comparison: Placebo vs TAK-063; PANSS Negative Score, Change at Week 2; Test type: Superiority or Other; p = 0.396, MMRM — No adjustment for multiple comparisons. Least square means, differences and p-values were obtained using a MMRM; MMRM = -0.59, 95% CI 2-sided [-1.96 to 0.78], Standard Error of Mean 0.693 — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 9: Comparison: Placebo vs TAK-063; PANSS Negative Score, Change at Week 3; Test type: Superiority or Other; p = 0.612, MMRM — No adjustment for multiple comparisons. Least square means, differences and p-values were obtained using a MMRM; Least square mean difference = -0.37, 95% CI 2-sided [-1.79 to 1.06], Standard Error of Mean 0.722 — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 10: Comparison: Placebo vs TAK-063; PANSS Negative Score, Change at Week 4; Test type: Superiority or Other; p = 0.670, MMRM — No adjustment for multiple comparisons. Least square means, differences and p-values were obtained using a MMRM; Least square mean difference = -0.37, 95% CI 2-sided [-2.06 to 1.33], Standard Error of Mean 0.856 — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 11: Comparison: Placebo vs TAK-063; PANSS Negative Score, Change at Week 5; Test type: Superiority or Other; p = 0.807, MMRM — No adjustment for multiple comparisons. Least square means, differences and p-values were obtained using a MMRM; Least square mean difference = -0.22, 95% CI 2-sided [-1.98 to 1.55], Standard Error of Mean 0.892 — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 12: Comparison: Placebo vs TAK-063; PANSS Negative Score, Change at Week 6; Test type: Superiority or Other; p = 0.182, MMRM — No adjustment for multiple comparisons. Least square means, differences and p-values were obtained using a MMRM; Least square mean difference = -1.14, 95% CI 2-sided [-2.83 to 0.54], Standard Error of Mean 0.853 — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 13: Comparison: Placebo vs TAK-063; PANSS General Score, Change at Week 1; Test type: Superiority or Other; p = 0.933, MMRM — No adjustment for multiple comparisons. Least square means, differences and p-values were obtained using a MMRM; Least square mean difference = 0.07, 95% CI 2-sided [-1.52 to 1.65], Standard Error of Mean 0.801 — TAK-063 - Placebo. PANSS subscale score as a covariate, pooled center, week and treatment as fixed factors, the treatment-by-week interaction and Baseline PANSS subscale score-by-week interaction
Statistical Analysis 14: Comparison: Placebo vs TAK-063; PANSS General Score, Change at Week 2; Test type: Superiority or Other; p = 0.596, MMRM — No adjustment for multiple comparisons. Least square means, differences and p-values were obtained using a MMRM; Least square mean difference = -0.61, 95% CI 2-sided [-2.89 to 1.66], Standard Error of Mean 1.151 — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 15: Comparison: Placebo vs TAK-063; PANSS General Score, Change at Week 3; Test type: Superiority or Other; p = 0.371, MMRM — No adjustment for multiple comparisons. Least square means, differences and p-values were obtained using a MMRM; Least square mean difference = -1.31, 95% CI 2-sided [-4.18 to 1.57], Standard Error of Mean 1.455 — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 16: Comparison: Placebo vs TAK-063; PANSS General Score, Change at Week 4; Test type: Superiority or Other; p = 0.821, MMRM — No adjustment for multiple comparisons. Least square means, differences and p-values were obtained using a MMRM; Least square mean difference = -0.37, 95% CI 2-sided [-3.58 to 2.84], Standard Error of Mean 1.625 — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 17: Comparison: Placebo vs TAK-063; PANSS General Score, Change at Week 5; Test type: Superiority or Other; p = 0.323, MMRM — No adjustment for multiple comparisons. Least square means, differences and p-values were obtained using a MMRM; Least square mean difference = -1.61, 95% CI 2-sided [-4.81 to 1.60], Standard Error of Mean 1.621 — [estimate comment as in outcome 4, analysis 13]
Statistical Analysis 18: Comparison: Placebo vs TAK-063; PANSS General Score, Change at Week 6; Test type: Superiority or Other; p = 0.161, MMRM — No adjustment for multiple comparisons. Least square means, differences and p-values were obtained using a MMRM; Least square mean difference = -2.44, 95% CI 2-sided [-5.87 to 0.98], Standard Error of Mean 1.732 — [estimate comment as in outcome 4, analysis 1]

5. Secondary Outcome: Percentage of Clinical Responders Based on the PANSS Total Score
Description: Clinical responders based on the PANSS total score is defined as at least 30% improvement from baseline in the total score. PANSS assesses the positive symptoms, negative symptoms, and general psychopathology specifically associated with schizophrenia. The scale consists of 30 items. Each item is rated on a scale from 1 (symptom not present) to 7 (symptoms extremely severe). The sum of the 30 items is defined as the PANSS total score and ranges from 30 to 210; higher score indicates greater severity.
Time Frame: Weeks 1, 2, 3, 4, 5 and 6
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | TAK-063
Number analyzed (Participants) | 76 | 80
percentage of participants
  Week 1 (n=76,80) | 6.6 | 20.0
  Week 2 (n=72,72) | 18.1 | 37.5
  Week 3 (n=67,68) | 26.9 | 39.7
  Week 4 (n=57,60) | 38.6 | 43.3
  Week 5 (n=53,58) | 37.7 | 48.3
  Week 6 (n=51,55) | 43.1 | 54.5
Statistical Analysis 1: Comparison: Placebo vs TAK-063; Week 1; Test type: Superiority or Other; p = 0.017, Regression, Logistic; Odds Ratio (OR) = 3.664, 95% CI 2-sided [1.263 to 10.624] — TAK-063 versus Placebo. The p-values were obtained using a logistic regression model adjusting for treatment and the Baseline PANSS total score
Statistical Analysis 2: Comparison: Placebo vs TAK-063; Week 2; Test type: Superiority or Other; p = 0.009, Regression, Logistic; Odds Ratio (OR) = 2.782, 95% CI 2-sided [1.287 to 6.014] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs TAK-063; Week 3; Test type: Superiority or Other; p = 0.108, Regression, Logistic; Odds Ratio (OR) = 1.818, 95% CI 2-sided [0.877 to 3.771] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 4: Comparison: Placebo vs TAK-063; Week 4; Test type: Superiority or Other; p = 0.596, Regression, Logistic; Odds Ratio (OR) = 1.222, 95% CI 2-sided [0.583 to 2.561] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 5: Comparison: Placebo vs TAK-063; Week 5; Test type: Superiority or Other; p = 0.263, Regression, Logistic; Odds Ratio (OR) = 1.542, 95% CI 2-sided [0.722 to 3.292] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 6: Comparison: Placebo vs TAK-063; Week 6; Test type: Superiority or Other; p = 0.253, Regression, Logistic; Odds Ratio (OR) = 1.567, 95% CI [0.725 to 3.388] — [estimate comment as in outcome 5, analysis 1]

6. Secondary Outcome: Change From Baseline in Clinical Global Impression - Severity (CGI-S) Score at Weeks 1, 2, 3, 4, 5,and 6
Description: The CGI-S is a clinician rated scale designed to assess global severity of illness. CGI-S is a 7-point scale that requires the clinician to rate the severity of the participant's illness at the time of assessment. A participant is assessed on severity of mental illness on the following scale: 1, normal, not at all ill; 2, borderline ill; 3, mildly ill; 4, moderately ill; 5, markedly ill; 6, severely ill; or 7, extremely ill. Least square mean and standard error values were determined using a MMRM. A negative change from Baseline indicates improvement.
Time Frame: Baseline, Weeks 1, 2, 3, 4, 5 and 6
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | TAK-063
Number analyzed (Participants) | 76 | 80
score on a scale
  Change at Week 1 (n=76,80) | -0.39 (0.069) | -0.44 (0.067)
  Change at Week 2 (n=72,72) | -0.45 (0.097) | -0.67 (0.096)
  Change at Week 3 (n=68,68) | -0.55 (0.118) | -0.99 (0.118)
  Change at Week 4 (n=57,60) | -0.58 (0.129) | -0.94 (0.127)
  Change at Week 5 (n=53,58) | -0.66 (0.137) | -1.13 (0.134)
  Change at Week 6 (n=51,55) | -0.76 (0.145) | -1.19 (0.141)
Statistical Analysis 1: Comparison: Placebo vs TAK-063; Change at Week 1; Test type: Superiority or Other; p = 0.619, MMRM — No adjustment for multiple comparisons. Least square means, differences and p-values were obtained using a MMRM; Least square mean difference = -0.05, 95% CI 2-sided [-0.23 to 0.14], Standard Error of Mean 0.095 — TAK-063 - Placebo. Baseline CGI-S score was used as a covariate, pooled center, week and treatment as fixed factors, the treatment-by-week interaction and Baseline CGI-S score-by-week interaction
Statistical Analysis 2: Comparison: Placebo vs TAK-063; Change at Week 2; Test type: Superiority or Other; p = 0.116, MMRM — No adjustment for multiple comparisons. Least square means, differences and p-values were obtained using a MMRM; Least square mean difference = -0.21, 95% CI 2-sided [-0.48 to 0.05], Standard Error of Mean 0.136 — [estimate comment as in outcome 6, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs TAK-063; Change at Week 3; Test type: Superiority or Other; p = 0.009, MMRM — No adjustment for multiple comparisons. Least square means, differences and p-values were obtained using a MMRM; Least square mean difference = -0.44, 95% CI 2-sided [-0.77 to -0.11], Standard Error of Mean 0.166 — [estimate comment as in outcome 6, analysis 1]
Statistical Analysis 4: Comparison: Placebo vs TAK-063; Change at Week 4; Test type: Superiority or Other; p = 0.049, MMRM — No adjustment for multiple comparisons. Least square means, differences and p-values were obtained using a MMRM; Least square mean difference = -0.36, 95% CI 2-sided [-0.72 to 0.00], Standard Error of Mean 0.180 — [estimate comment as in outcome 6, analysis 1]
Statistical Analysis 5: Comparison: Placebo vs TAK-063; Change at Week 5; Test type: Superiority or Other; p = 0.016, MMRM — No adjustment for multiple comparisons. Least square means, differences and p-values were obtained using a MMRM; Least square mean difference = -0.47, 95% CI 2-sided [-0.85 to -0.09], Standard Error of Mean 0.191 — [estimate comment as in outcome 6, analysis 1]
Statistical Analysis 6: Comparison: Placebo vs TAK-063; Change at Week 6; Test type: Superiority or Other; p = 0.035, MMRM — No adjustment for multiple comparisons. Least square means, differences and p-values were obtained using a MMRM; Least square mean difference = -0.43, 95% CI [-0.83 to -0.03], Standard Error of Mean 0.202 — [estimate comment as in outcome 6, analysis 1]

7. Secondary Outcome: Clinical Global Impression Scale - Improvement (CGI-I) Score at Weeks 1, 2, 3, 4, 5 and 6
Description: The CGI-I assesses the participant's improvement (or worsening). The clinician is required to assess the participant's condition relative to baseline on a 7-point scale. CGI-I scale assesses the participant's improvement (or worsening) on a 7-point scale: 1, very much improved; 2, much improved; 3, minimally improved; 4, no change; 5, minimally worse; 6, much worse; or 7, very much worse. Least square mean and standard error values were calculated using a MMRM.
Time Frame: Weeks 1, 2, 3, 4, 5 and 6
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | TAK-063
Number analyzed (Participants) | 76 | 80
score on a scale
  Week 1 (n=76,80) | 3.53 (0.093) | 3.49 (0.091)
  Week 2 (n=72,72) | 3.58 (0.124) | 3.20 (0.123)
  Week 3 (n=67,68) | 3.63 (0.144) | 3.07 (0.144)
  Week 4 (n=57,60) | 3.53 (0.157) | 2.97 (0.155)
  Week 5 (n=53,58) | 3.54 (0.171) | 2.98 (0.167)
  Week 6 (n=51,55) | 3.46 (0.175) | 2.80 (0.171)
Statistical Analysis 1: Comparison: Placebo vs TAK-063; Week 1; Test type: Superiority or Other; p = 0.746, MMRM — No adjustment for multiple comparisons. Least square means, differences and p-values were obtained using a MMRM; Least square mean difference = -0.04, 95% CI 2-sided [-0.29 to 0.21], Standard Error of Mean 0.128 — [estimate comment as in outcome 6, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs TAK-063; Week 2; Test type: Superiority or Other; p = 0.034, MMRM — No adjustment for multiple comparisons. Least square means, differences and p-values were obtained using a MMRM; Least mean square difference = -0.37, 95% CI 2-sided [-0.72 to -0.03], Standard Error of Mean 0.173 — [estimate comment as in outcome 6, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs TAK-063; Week 3; Test type: Superiority or Other; p = 0.006, MMRM — No adjustment for multiple comparisons. Least square means, differences and p-values were obtained using a MMRM; Least square mean difference = -0.57, 95% CI 2-sided [-0.97 to -0.17], Standard Error of Mean 0.203 — [estimate comment as in outcome 6, analysis 1]
Statistical Analysis 4: Comparison: Placebo vs TAK-063; Week 4; Test type: Superiority or Other; p = 0.013, MMRM — No adjustment for multiple comparisons. Least square means, differences and p-values were obtained using a MMRM; Least square mean difference = -0.55, 95% CI 2-sided [-0.99 to -0.12], Standard Error of Mean 0.220 — [estimate comment as in outcome 6, analysis 1]
Statistical Analysis 5: Comparison: Placebo vs TAK-063; Week 5; Test type: Superiority or Other; p = 0.020, MMRM — No adjustment for multiple comparisons. Least square means, differences and p-values were obtained using a MMRM; Least mean square difference = -0.56, 95% CI 2-sided [-1.03 to -0.09], Standard Error of Mean 0.238 — [estimate comment as in outcome 6, analysis 1]
Statistical Analysis 6: Comparison: Placebo vs TAK-063; Week 6; Test type: Superiority or Other; p = 0.007, MMRM — No adjustment for multiple comparisons. Least square means, differences and p-values were obtained using a MMRM; Least square mean difference = -0.66, 95% CI 2-sided [-1.15 to -0.18], Standard Error of Mean 0.244 — [estimate comment as in outcome 6, analysis 1]

8. Secondary Outcome: Percentage of Responders Based on CGI-I Ratings Score
Description: Responder based on CGI-I is defined as a rating of much improved or very much improved. The CGI-I assesses the participant's improvement (or worsening). The clinician is required to assess the participant's condition relative to baseline on a 7-point scale: 1, very much improved; 2, much improved; 3, minimally improved; 4, no change; 5, minimally worse; 6, much worse; or 7, very much worse.
Time Frame: Weeks 1, 2, 3, 4, 5 and 6
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | TAK-063
Number analyzed (Participants) | 76 | 80
percentage of participants
  Week 1 (n=76,80) | 6.6 | 15.0
  Week 2 (n=72,72) | 18.1 | 31.9
  Week 3 (n=67,68) | 19.4 | 36.8
  Week 4 (n=57,60) | 31.6 | 43.3
  Week 5 (n=53,58) | 32.1 | 44.8
  Week 6 (n=51,55) | 29.4 | 58.2
Statistical Analysis 1: Comparison: Placebo vs TAK-063; Week 1; Test type: Superiority or Other; p = 0.077, Regression, Logistic — No multiplicity adjustment; Odds Ratio (OR) = 2.726, 95% CI 2-sided [0.899 to 8.267] — TAK-063 versus Placebo. The p-values were obtained using a logistic regression model adjusting for treatment and the Baseline CGI-S score
Statistical Analysis 2: Comparison: Placebo vs TAK-063; Week 2; Test type: Superiority or Other; p = 0.036, Regression, Logistic — No multiplicity adjustment; Odds Ratio (OR) = 2.331, 95% CI 2-sided [1.055 to 5.153] — [estimate comment as in outcome 8, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs TAK-063; Week 3; Test type: Superiority or Other; p = 0.015, Regression, Logistic — No multiplicity adjustment; Odds Ratio (OR) = 2.690, 95% CI 2-sided [1.208 to 5.990] — [estimate comment as in outcome 8, analysis 1]
Statistical Analysis 4: Comparison: Placebo vs TAK-063; Week 4; Test type: Superiority or Other; p = 0.158, Regression, Logistic — No multiplicity adjustment; Odds Ratio (OR) = 1.737, 95% CI 2-sided [0.807 to 3.735] — [estimate comment as in outcome 8, analysis 1]
Statistical Analysis 5: Comparison: Placebo vs TAK-063; Week 5; Test type: Superiority or Other; p = 0.164, Regression, Logistic — No multiplicity adjustment; Odds Ratio (OR) = 1.739, 95% CI 2-sided [0.798 to 3.789] — [estimate comment as in outcome 8, analysis 1]
Statistical Analysis 6: Comparison: Placebo vs TAK-063; Week 6; Test type: Superiority or Other; p = 0.003, Regression, Logistic — No multiplicity adjustment; Odds Ratio (OR) = 3.440, 95% CI 2-sided [1.523 to 7.770] — [estimate comment as in outcome 8, analysis 1]

9. Secondary Outcome: Change From Baseline in Brief Assessment of Cognition in Schizophrenia (BACS) Score at Weeks 3 and 6
Description: BACS is specifically designed to measure treatment- related improvements in cognition and includes alternate forms. The battery of tests in the BACS includes brief assessments of reasoning and problem solving, verbal fluency, attention, verbal memory, working memory, and motor speed. The primary measure from each test of the BACS is standardized by creating z-scores whereby the mean of the test session of a healthy participant is set to 0 and the standard deviation set to 1. A composite score was calculated by averaging all of the 6 standardized primary measures from the BACS, and then calculating a z-score of the composite. The composite z-score indicates how much higher or lower the participant's cognition is compared to a healthy person. Least square mean and standard error values were determined using a MMRM.
Time Frame: Baseline, Weeks 3 and 6
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: z-score
Arm/Group | Placebo | TAK-063
Number analyzed (Participants) | 76 | 80
z-score
  Change at Week 3 (n=69,71) | 0.69 (1.120) | 2.49 (1.104)
  Change at Week 6 (n=49,54) | 2.33 (1.290) | 4.52 (1.251)
Statistical Analysis 1: Comparison: Placebo vs TAK-063; Change at Week 3; Test type: Superiority or Other; p = 0.246, MMRM — No adjustment for multiple comparisons. Least square means, differences and p-values were obtained using a MMRM; Least square mean difference = 1.80, 95% CI 2-sided [-1.26 to 4.86], Standard Error of Mean 1.547 — TAK-063 - Placebo. Baseline BACS total score was used as a covariate, pooled center, week and treatment as fixed factors, the treatment-by-week interaction and Baseline BACS total score-by-week interaction
Statistical Analysis 2: Comparison: Placebo vs TAK-063; Change at Week 6; Test type: Superiority or Other; p = 0.216, Least square mean difference — No adjustment for multiple comparisons. Least square means, differences and p-values were obtained using a MMRM; Least square mean difference = 2.20, 95% CI 2-sided [-1.30 to 5.69], Standard Error of Mean 1.767 — [estimate comment as in outcome 9, analysis 1]

10. Secondary Outcome: Change From Baseline in Brief Negative Symptom Scale (BNSS) Score at Weeks 3 and 6
Description: The BNSS is a13-item instrument designed for use in clinical trials and other studies that measures 5 domains of negative symptoms: blunted affect, alogia, asociality, anhedonia, and avolition. All the items in the BNSS are rated on a 7-point (0-6) scale, with anchor points generally ranging from the symptom's being absent (0) to severe (6). A scale total score is calculated by summing the 13 individual items; total score range of 0 to 78, where higher score indicates higher severity of negative symptoms. Least square mean and standard error values were determined using a MMRM. A negative change from Baseline indicates improvement.
Time Frame: Baseline, Weeks 3 and 6
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | TAK-063
Number analyzed (Participants) | 76 | 80
score on a scale
  Change at Week 3 (n=71,75) | -3.70 (1.217) | -4.08 (1.185)
  Change at Week 6 (n=51,55) | -4.93 (1.498) | -7.80 (1.451)
Statistical Analysis 1: Comparison: Placebo vs TAK-063; Change at Week 3; Test type: Superiority or Other; p = 0.820, MMRM — No adjustment for multiple comparisons. Least square means, differences and p-values were obtained using a MMRM; Least mean square difference = -0.38, 95% CI 2-sided [-3.67 to 2.91], Standard Error of Mean 1.664 — TAK-063 - Placebo. Baseline BNSS total score was used as a covariate, pooled center, week and treatment as fixed factors, the treatment-by-week interaction and Baseline BNSS total score-by-week interaction
Statistical Analysis 2: Comparison: Placebo vs TAK-063; Change at Week 6; Test type: Superiority or Other; p = 0.163, MMRM — No adjustment for multiple comparisons. Least square means, differences and p-values were obtained using a MMRM; Least square mean difference = -2.87, 95% CI 2-sided [-6.93 to 1.18], Standard Error of Mean 2.050 — TAK-063 - Placebo. Baseline BNSS total score was used as a covariate, pooled center, week and treatment as fixed factors, the treatment-by-week interaction and Baseline BACS total score-by-week interaction

11. Secondary Outcome: Change From Baseline in the Personal and Social Performance (PSP) Scale Score at Weeks 3 and 6
Description: The PSP scale is a clinician-reported outcome instrument that was developed to evaluate social and personal functioning. It measures 4 domains of social functioning: socially useful activities including work and study, personal and social relationships, self-care and disturbing and aggressive behaviors. The clinician assigns an initial 6-degree of severity to each area (absent, mild, manifest, marked, severe or very severe). The final result is a single assessment of social functioning ranging from 0 (no autonomy) to 100 (excellent functioning). Least square mean and standard error values were determined using a MMRM. A positive change from Baseline indicates improvement.
Time Frame: Baseline, Weeks 3 and 6
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | TAK-063
Number analyzed (Participants) | 76 | 80
score on a scale
  Change at Week 3 (n=70,75) | 7.19 (1.301) | 9.88 (1.244)
  Change at Week 6 (n=50,55) | 9.65 (1.693) | 12.27 (1.605)
Statistical Analysis 1: Comparison: Placebo vs TAK-063; Change at Week 3; Test type: Superiority or Other; p = 0.131, MMRM — No adjustment for multiple comparisons. Least square means, differences and p-values were obtained using a MMRM; Least square mean difference = 2.69, 95% CI 2-sided [-0.81 to 6.19], Standard Error of Mean 1.769 — TAK-063 - Placebo. Baseline PSP score was used as a covariate, pooled center, week and treatment as fixed factors, the treatment-by-week interaction and Baseline PSP score-by-week interaction
Statistical Analysis 2: Comparison: Placebo vs TAK-063; Change at Week 6; Test type: Superiority or Other; p = 0.260, MMRM — No adjustment for multiple comparisons. Least square means, differences and p-values were obtained using a MMRM; Least square mean difference = 2.62, 95% CI 2-sided [-1.96 to 7.19], Standard Error of Mean 2.313 — [estimate comment as in outcome 11, analysis 1]

12. Secondary Outcome: Change From Baseline in the University of California San Diego Performance-based Skills Assessment - Brief Version (UPSA-B) at Week 3 and 6
Description: The UPSA-B evaluates the abilities of individuals to perform everyday tasks that are considered necessary for independent functioning in the community. The UPSA-B uses role playing situations to evaluate skills in 5 areas: household chores, communication, finance, transportation, and planning recreational activities. Subscale scores range from 0 to 20 points, and total scores range from 0 to 100 points; higher scores reflect better performance. Least square mean and standard error values were determined using a MMRM. A positive change from Baseline indicates improvement.
Time Frame: Baseline, Weeks 3 and 6
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | TAK-063
Number analyzed (Participants) | 76 | 80
score on a scale
  Change at Week 3 (n=69,71) | 2.13 (1.337) | 2.20 (1.322)
  Change at Week 6 (n=49,54) | 3.97 (1.656) | 3.43 (1.592)
Statistical Analysis 1: Comparison: Placebo vs TAK-063; Change at Week 3; Test type: Superiority or Other; p = 0.973, MMRM — No adjustment for multiple comparisons. Least square means, differences and p-values were obtained using a MMRM; Least square mean difference = 0.06, 95% CI 2-sided [-3.61 to 3.73], Standard Error of Mean 1.855 — TAK-063 - Placebo. Baseline UPSA-B composite score was used as a covariate, pooled center, week and treatment as fixed factors, the treatment-by-week interaction and Baseline UPSA-B composite score-by-week interaction
Statistical Analysis 2: Comparison: Placebo vs TAK-063; Change at Week 6; Test type: Superiority or Other; p = 0.812, MMRM — No adjustment for multiple comparisons. Least square means, differences and p-values were obtained using a MMRM; Least mean square difference = -0.54, 95% CI 2-sided [-5.00 to 3.92], Standard Error of Mean 2.255 — [estimate comment as in outcome 12, analysis 1]

ADVERSE EVENTS:
Time Frame: Up to 14 days after the last dose (Up to Week 8)
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Placebo | TAK-063
Serious Adverse Events (participants affected / at risk) | 2/81 | 4/83
Other Adverse Events (participants affected / at risk) | 42/81 | 58/83
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=81) | TAK-063 (N=83)
Cellulitis (Infections and infestations) | 1 | 0
Agitation (Psychiatric disorders) | 1 | 1
Schizophrenia (Psychiatric disorders) | 0 | 2
Suicidal ideation (Psychiatric disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=81) | TAK-063 (N=83)
Dyspepsia (Gastrointestinal disorders) | 6 | 9
Nausea (Gastrointestinal disorders) | 5 | 5
Constipation (Gastrointestinal disorders) | 6 | 3
Neck pain (Musculoskeletal and connective tissue disorders) | 6 | 1
Akathisia (Nervous system disorders) | 4 | 11
Headache (Nervous system disorders) | 9 | 6
Somnolence (Nervous system disorders) | 2 | 10
Dystonia (Nervous system disorders) | 1 | 5
Decreased appetite (Metabolism and nutrition disorders) | 1 | 5
Toothache (Gastrointestinal disorders) | 2 | 4
Vomiting (Gastrointestinal disorders) | 2 | 4
Dry mouth (Gastrointestinal disorders) | 3 | 2
Diarrhoea (Gastrointestinal disorders) | 1 | 3
Abdominal discomfort (Gastrointestinal disorders) | 3 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 2
Abdominal pain upper (Gastrointestinal disorders) | 1 | 2
Pain (General disorders) | 2 | 1
Nasopharyngitis (Infections and infestations) | 1 | 2
Tooth abscess (Infections and infestations) | 1 | 2
Upper respiratory tract infection (Infections and infestations) | 2 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 3
Weight increased (Investigations) | 3 | 2
Increased appetite (Metabolism and nutrition disorders) | 2 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 4 | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 2
Torticollis (Musculoskeletal and connective tissue disorders) | 0 | 2
Trismus (Musculoskeletal and connective tissue disorders) | 0 | 2
Dizziness (Nervous system disorders) | 3 | 1
Paraesthesia (Nervous system disorders) | 1 | 2
Tremor (Nervous system disorders) | 2 | 1
Anxiety (Psychiatric disorders) | 1 | 3
Insomnia (Psychiatric disorders) | 3 | 0
Psychotic disorder (Psychiatric disorders) | 1 | 2
Agitation (Psychiatric disorders) | 2 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Hot flush (Vascular disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.